CLINICAL TRIAL: NCT05224765
Title: Reducing G60 Recidivism Rates
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 036.TRA.2021.A
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Fall Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Geriatric patients that attended fall prevention discharge class: recidivism rates of MDMC-qualified G60 patients that attended fall prevention discharge class per hospital protocols
  Interventions: Other: Fall prevention class
- Geriatric patients that did not attend fall prevention discharge class: recidivism rates of MDMC-qualified G60 patients that did not attended fall prevention discharge class per hospital protocols

INTERVENTIONS:
Other: Fall prevention class — Participants attend fall prevention discharge class per hospital protocols
  Groups: Geriatric patients that attended fall prevention discharge class

SUMMARY:
The research surrounding best practice guidelines of geriatric trauma patients in the inpatient setting is broad. Furthermore, the comprehensiveness of research programs varies based on individual hospital resource capacity. American College of Surgeons Trauma Quality Improvement Program (ACS TQIP) Geriatric Trauma Management Guidelines1 details a comprehensive, multidisciplinary approach to inpatient management; however, guideline effectiveness is diminished as many hospitals may implement a version of the guidelines limited by staffing, ancillary services, and resource capacity, among other variables.

DETAILED DESCRIPTION:
Risk of future falls in elderly patients increases based on multiple factors including increased age and history of previous falls. However, there is limited research showing evidenced-based interventions that reduce recidivism rates related to falls. The Centers for Disease Control and Prevention (CDC) has an evidenced-based fall prevention program (Stopping Elderly Accidents, Deaths & Injuries [STEADI3]). Implementation of STEADI as part of a multidisciplinary approach to fall risk assessment and prevention prior to discharge may reduce recidivism in elderly patients.

Ground level falls are the most common mechanism of injury in older adults and are increasingly becoming a significant cause of morbidity and mortality in this population. An individual's risk of a repeat ground level fall increases after an initial fall, injury, or hospitalization7. Addressing fall risk factors and tailoring inpatient care for any trauma in the elderly population prior to discharge will likely improve outcomes, decrease length of stay, and decrease morbidity and mortality.

The introduction of STEADI as part of a specialized multidisciplinary approach to fall risk assessment and prevention prior to hospital discharge may reduce recidivism in elderly patients. Patients that attend the discharge class are typically more likely to go home and return to independence whereas those that do not attend the discharge class are likely to have a disposition of going to a long-term care facility or are not mentally capable of retaining information. Reduced falls as a result of STEADI implementation will putatively improve mortality rates and quality of life in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* G60 activation and admission
* Primary admission for injury

Exclusion Criteria:

* Less than 60 years old
* Admitted for non-traumatic injuries
* Non-index admission for injury
* Prisoners
* Pregnant or lactating subjects

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: G60 patients across all MHS hospitals between 2019 and 2022
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with repeat ED visits with a chief complaint associated with a fall. | 2019-2022
  review of G60 patients across all MHS hospitals after system standard order set initiation and utilization as the comparative group for a 2-year period.
• Number of return visits related to a fall treated at a MHS trauma center before and after implementation of G60 targeted education. | 2019-2022
  • Observational study comparing recidivism rates of MDMC-qualified G60 patients that attended fall prevention discharge class per hospital protocols versus G60 patients that did not attend the class

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bradley, RN, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States